CLINICAL TRIAL: NCT00911300
Title: An International, Multicentre, Randomised, Open, Controlled, Two-parallel Group, Phase II Pilot Study to Evaluate the Efficacy and Safety of ARIXTRA™ for Anticoagulation of Patients With Atrial Fibrillation Undergoing Electric Cardioversion Following Transesophageal Echocardiography
Brief Title: Evaluation of Fondaparinux in Patients With a Heart Rhythm Disturbance Who Undergo Restoration of Normal Heart Rhythm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111418
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Fibrillation, Atrial
Keywords: Cardioversion, Electric; Pathological Conditions, Sings and Symptoms; Cardiovascular Diseases; Heart Diseases; Atrial Fibrillation; Arrhythmias, Cardiac; Pathologic Processes; Anticoagulants
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases; Heart Diseases; Arrhythmias, Cardiac; Pathologic Processes | interventions — Fondaparinux; Heparin; acarboxyprothrombin

ARMS (2):
- Arm 1: fondaparinux (Active Comparator)
  Interventions: Drug: fondaparinux
- Arm 2: unfractionated heparin + Vitamin-K-Antagonist (Active Comparator)
  Interventions: Drug: unfractionated heparin; Drug: Vitamin-K-Antagonist

INTERVENTIONS:
Drug: fondaparinux — Comparison of different drugs
  Arms: Arm 1: fondaparinux
Drug: unfractionated heparin — Comparison of different drugs
  Arms: Arm 2: unfractionated heparin + Vitamin-K-Antagonist
Drug: Vitamin-K-Antagonist — Comparison of different drugs
  Arms: Arm 2: unfractionated heparin + Vitamin-K-Antagonist

SUMMARY:
The purpose of this study is to test whether Fondaparinux is effective and safe to prevent thromboembolic events (like for example strokes) and bleeding events in patients who undergo a normalisation of their heart rhythm disturbance. Fondaparinux will be compared with Heparin and tablets containing Vitamin-K-Antagonists (Phenprocoumon, Fluindione, or Warfarin).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged at least 18 years with atrial fibrillation (AF) meeting at least one of the following criteria (a, b, c): a. Acute clinical symptoms (like palpitations, chest pain, dyspnea, fatigue, lightheadedness, or syncope) for at least 48 hours and AF on baseline ECG b. Newly discovered AF persisting for >=7 days c. Recurrent AF persisting for >=7 days

Exclusion Criteria:

* No documented sinus rhythm on ECG for more than 1 year
* Acute neurological deficits (TIA, stroke, intracranial bleeding), or known disease which may cause neurological deficits (e.g., multiple sclerosis, seizure disorder)
* Treatment with antithrombotic agents, including low-dose anticoagulation, for more than 48 hours prior to randomisation
* Treatment with oral NSAIDs or ASA at doses greater than 325 mg per day for more than 72 hours prior to randomisation
* Anticoagulant therapy required or likely to be required during the study period
* Treatment with ASA at a dose greater than 325 mg per day or oral NSAIDs (at any dose) required or likely to be required during the study period
* Treatment with two or more antiplatelet agents (e.g. clopidogrel and ASA) at any dose at the same time (i.e., within 24 hours)
* Known hypersensitivity to UFH, VKA, or Fondaparinux or one of these drugs' excipients
* Active, clinically significant bleeding or clinically significant bleeding within the past month
* Major surgery within the previous three months
* Uncontrolled arterial hypertension (persistent systolic blood pressure over 180 mm Hg or diastolic blood pressure over 110 mm Hg)
* Bacterial endocarditis
* Calculated creatinine clearance < 30 mL/min
* Body weight < 50 kg
* Planned surgery or intervention within the next 65 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- France (12):
  - GSK Investigational Site, Albi
  - GSK Investigational Site, Antony
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Évecquemont
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pau
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Toulouse
- Germany (16):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Bad Tölz, Bavaria
  - GSK Investigational Site, Simbach A. Inn, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Hagenow, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg-Huckingen, North Rhine-Westphalia
  - GSK Investigational Site, Unna, North Rhine-Westphalia
  - GSK Investigational Site, Wesel, North Rhine-Westphalia
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) were required to undergo transesophageal echocardiography (TEE) to guide cardioversion (CV). TEEs were recorded and archived to allow for later central adjudication and possible evaluation of details. At randomization (Day 1, immediately after TEE), par. were stratified to thrombus (clot)-positive and thrombus (clot)-negative.
Groups:
- Fondaparinux: For clot-negative (CN) participants (par.), 7.5 milligrams (mg) fondaparinux was injected once daily (OD) subcutaneously (for par. with body weight [BW] 50-100 kilograms [kg]); for par. with BW >100 kg, 10 mg fondaparinux was administered using a disposable prefilled syringe for the first 7-10 days after randomization, followed by 3 weeks of 2.5 mg fondaparinux OD (until Day 28+/-4). For clot-positive (CP) par. with creatinine clearance (CrCl) >= 50 milliliters (mL)/minute (min), 7.5 mg fondaparinux was injected OD (for par. with BW 50-100 kg); for par. with BW >100 kg, 10 mg fondaparinux was administered OD. For CP par. with CrCl 30 to <50 mL/min, 5 mg fondaparinux was injected OD (for par. with BW 50-100 kg); for par. with BW >100 kg, 7.5 mg fondaparinux was injected for 28+/-4 days. If the second TEE showed thrombus disappearance, treatment continued until 7-10 days after the second TEE followed by 3 weeks of 2.5 mg fondaparinux OD (total treatment duration: 56+/-4 days).
- Unfractioned Heparin (UFH)/Vitamin K Antagonist (VKA): Both CN and CP participants received an initial intravenous (i.v.) bolus injection of 70 international units (IU)/kg (at least 5000 IU) UFH, followed by continuous infusion at an initial rate of 15 IU/kg/hour (h) (at least 1250 IU per hour). The infusion dose was adjusted to maintain an activated partial thromboplastin time (aPTT) at 1.5 to 2 times the reference control value. Infusion continued for at least 72 h. In parallel to UFH, treatment with VKA was started as soon as possible (preferably on Day 1). The dose of VKA was adjusted to reach a target international normalized ratio (INR) of 2.0-3.0. UFH was continued until INR >2.0. Total treatment duration: 28+/-4 days. For CP participants for whom the second TEE showed thrombus disappearance, VKA was continued during cardioversion and up to a total treatment duration of 56+/-4 days.
Period: Overall Study
Arm/Group | Fondaparinux | Unfractioned Heparin (UFH)/Vitamin K Antagonist (VKA)
Started | 175 | 174
Completed | 140 | 131
Not Completed | 35 | 43
Not completed — Primary Endpoint Component Occurred | 1 | 2
Not completed — Death | 1 | 0
Not completed — Thrombus Persistant in Second TEE | 3 | 7
Not completed — Adverse Event | 14 | 6
Not completed — Protocol Violation | 3 | 2
Not completed — Consent Withdrawn | 4 | 12
Not completed — Coronary Angiography Performed | 1 | 0
Not completed — Atrial Fibrillation (AF) Recurrence | 3 | 3
Not completed — Received Commercial Treatment | 1 | 0
Not completed — Recurrent Tachyarrhythmia | 1 | 1
Not completed — Recurrent Tachy-Arrhythmia Absoluta | 1 | 1
Not completed — Nurse Unavailable in Participant's City | 1 | 0
Not completed — CV Unsuccessful; Phenprocoumon Received | 1 | 0
Not completed — Participant Could Not Stay in Hospital | 0 | 1
Not completed — Investigator's Decision; New AF Episode | 0 | 1
Not completed — International Normalized Ratio Too High | 0 | 1
Not completed — Participant Refused Hospital Consulation | 0 | 1
Not completed — Underlying Disease (Myocarditis) | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Treatment Stopped by Mistake | 0 | 1
Not completed — Randomized; No Study Medication Received | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Fondaparinux: For CN par., 7.5 mg fondaparinux was injected OD subcutaneously (for par. with BW 50-100 kg; for par. with BW >100 kg, 10 mg fondaparinux was administered using a disposable prefilled syringe for the first 7-10 days after randomization, followed by 3 weeks of 2.5 mg fondaparinux OD (until Day 28+/-4). For CP par. with CrCl >= 50 mL/min, 7.5 mg fondaparinux was injected OD (for par. with BW 50-100 kg); for par. with BW >100 kg, 10 mg fondaparinux was administered OD. For CP par. with CrCl 30 to <50 mL/min, 5 mg fondaparinux was injected OD (for par. with BW 50-100 kg); for par. with BW >100 kg, 7.5 mg fondaparinux was injected for 28+/-4 days. If the second TEE showed thrombus disappearance, treatment continued until 7-10 days after the second TEE followed by 3 weeks of 2.5 mg fondaparinux OD (total treatment duration: 56+/-4 days).
- UFH/VKA: Both CN and CP participants received an initial i.v. bolus injection of 70 IU/kg (at least 5000 IU) UFH, followed by continuous infusion at an initial rate of 15 IU/kg/h (at least 1250 IU per h). The infusion dose was adjusted to maintain an activated partial thromboplastin aPTT at 1.5 to 2 times the reference control value. Infusion continued for at least 72 h. In parallel to UFH, treatment with VKA was started as soon as possible (preferably on Day 1). The dose of VKA was adjusted to reach a target INR of 2.0-3.0. UFH was continued until INR >2.0. Total treatment duration: 28+/-4 days. For CP participants for whom the second TEE showed thrombus disappearance, VKA was continued during cardioversion and up to a total treatment duration of 56+/-4 days.
- Total: Total of all reporting groups
Arm/Group | Fondaparinux | UFH/VKA | Total
Number analyzed (Participants) | 174 | 170 | 344
Age Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristic data were collected in members of the Modified Intent-to-Treat (mITT) Population, comprised of all randomized participants receiving at least one dose of study medication and for whom any post-baseline value was available.
  Years | 68.24 (11.09) | 66.78 (11.93) | 67.52 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristic data were collected in members of the Modified Intent-to-Treat (mITT) Population, comprised of all randomized participants receiving at least one dose of study medication and for whom any post-baseline value was available.
  Participants
    Female | 69 | 60 | 129
    Male | 105 | 110 | 215

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Event of Cerebral Neurologic Event, Systemic Thromboembolism, Death From Any Cause, and/or Major Bleeding Until the End of Treatment (EOT) Plus 4 Days
Description: Cerebral neurologic events are defined as any new neurologic disorders caused by cerebrovascular embolization, e.g., Transient Ischemic Attack (TIA), cerebral infarction. The cerebrovascular origin of the event has to be confirmed by objective procedures. Systemic thromboembolism comprises any arterial thromboembolic event (e.g., peripheral vascular embolism, mesenteric infarct, or myocardial infarction). All cerebral neurologic events were adjudicated by a Central Adjudication Committee (CAC), members of which were unaware of the participants' treatment assignment.
Time Frame: Baseline (Day 1) until Day 64 (4 days after the EOT [i.e., last administration of study drug]) for CP participants; Baseline until Day 36 (4 days after the EOT) for CN participants
Population: Modified Intent-to-Treat (mITT) Population: all randomized participants receiving at least one dose of study medication and for whom any post-baseline value was available
Measure: Number; unit: participants
Arm/Group | Fondaparinux | UFH/VKA
Number analyzed (Participants) | 174 | 170
participants | 3 | 2
Statistical Analysis 1: Comparison: Fondaparinux vs UFH/VKA; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percentage of participants = 0.5, 95% CI 2-sided [-2.0 to 3.1] — The estimated value is the absolute percent difference between Fondaparinux and UFH/VKA

2. Secondary Outcome: Number of Thrombus-negative and Thrombus-positive Participants (Par.) With at Least One Cerebral Neurologic Event
Description: Cerebral neurologic events are defined as any new neurologic disorders caused by cerebrovascular embolisation, e.g., TIA, cerebral infarction. All cerebral neurologic events were adjudicated by a CAC, members of which were unaware of the participants' treatment assignment.The cerebrovascular origin of the event was confirmed by objective procedures. A thrombus or blood clot is the final product of the blood coagulation step in hemostasis. It is achieved via the aggregation of platelets that form a platelet plug, and the activation of the humoral coagulation system (i.e., clotting factors).
Time Frame: Baseline (Day 1) until Day 64 (4 days after the EOT [i.e., last administration of study drug]) for CP participants; Baseline until Day 36 (4 days after the EOT) for CN participants; and from Baseline until the follow-up visit (FU) (Day 90+/-7)
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Fondaparinux | UFH/VKA
Number analyzed (Participants) | 174 | 170
participants
  Thrombus-negative par. until 4 days after EOT | 0 | 1
  Thrombus-positive par. until 4 days after EOT | 0 | 0
  Thrombus-negative participants until the FU | 1 | 1
  Thrombus-positive participants until the FU | 0 | 0

3. Secondary Outcome: Number of Thrombus-negative and Thrombus-positive Participants With at Least One Systemic Thromboembolism
Description: Systemic thromboembolism comprises any arterial thromboembolic event (e.g., peripheral vascular embolism, mesenteric infarct, or myocardial infarction). All systemic thromboembolic events were adjudicated by a CAC, the members of which were unaware of the participants' treatment assignment. A thrombus or blood clot is the final product of the blood coagulation step in hemostasis. It is achieved via the aggregation of platelets that form a platelet plug, and the activation of the humoral coagulation system (i.e., clotting factors).
Time Frame: as for outcome 2
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Fondaparinux | UFH/VKA
Number analyzed (Participants) | 174 | 170
participants
  Thrombus-negative par. until 4 days after EOT | 0 | 0
  Thrombus-positive par. until 4 days after EOT | 0 | 0
  Thrombus-negative participants until the FU | 0 | 0
  Thrombus-positive participants until the FU | 0 | 0

4. Secondary Outcome: Number of Thrombus-negative and Thrombus-positive Participants Who Died From Any Cause
Description: The cause of death was classified as due to a thromboembolic event (like cerebral infarction), bleeding, or other established diagnosis, or as unexplained. All deaths were adjudicated by an independent CAC, the members of which were unaware of the participants' treatment assignment. A thrombus or blood clot is the final product of the blood coagulation step in hemostasis. It is achieved via the aggregation of platelets that form a platelet plug, and the activation of the humoral coagulation system (i.e., clotting factors).
Time Frame: as for outcome 2
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Fondaparinux | UFH/VKA
Number analyzed (Participants) | 174 | 170
participants
  Thrombus-negative par. until 4 days after EOT | 1 | 0
  Thrombus-positive par. until 4 days after EOT | 0 | 0
  Thrombus-negative participants until the FU | 3 | 0
  Thrombus-positive participants until the FU | 0 | 0

5. Secondary Outcome: Number of Thrombus-negative and Thrombus-positive Participants With at Least One Major Bleeding Event
Description: Major bleeding: fatal, and/or symptomatic in a critical area/ organ, causes a fall in hemoglobin of >=3 grams/deciliter compared with the pre-randomization level, or leads to the transfusion of >=2 units of whole blood/red blood cells. All bleeding events were adjudicated by a CAC, the members of which were unaware of the participants' treatment assignment. A thrombus/ blood clot is the final product of the blood coagulation step in hemostasis. It is achieved via the aggregation of platelets, and the activation of the humoral coagulation system (i.e., clotting factors).
Time Frame: as for outcome 2
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Fondaparinux | UFH/VKA
Number analyzed (Participants) | 174 | 170
participants
  Thrombus-negative par. until 4 days after EOT | 3 | 1
  Thrombus-positive par. until 4 days after EOT | 0 | 0
  Thrombus-negative participants until the FU | 4 | 1
  Thrombus-positive participants until the FU | 0 | 0

6. Secondary Outcome: Number of Thrombus-negative and Thrombus-positive Participants With at Least One Minor Bleeding Event
Description: Minor bleeding is defined as clinically overt bleeding events that do not meet the criteria for major or clinically relevant non-major bleeding. All episodes of bleeding were adjudicated by an independent CAC, the members of which were unaware of the participants' treatment assignment.
Time Frame: as for outcome 2
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Fondaparinux | UFH/VKA
Number analyzed (Participants) | 174 | 170
participants
  Thrombus-negative par. until 4 days after EOT | 3 | 4
  Thrombus-positive par. until 4 days after EOT | 0 | 0
  Thrombus-negative participants until the FU | 3 | 5
  Thrombus-positive participants until the FU | 1 | 0

7. Secondary Outcome: Number of Participants With Primary Successful Electrical Cardioversion (CV) in Sinus Rhythm
Description: CV may be performed electively to restore sinus rhythm in patients with persistent AF. The primary successful electric CV was assessed by a 12- lead electrocardiogram (ECG) directly after the CV. Results of the last cardioversion were used in cases for which more than one CV was performed.
Time Frame: Day 1 until Day 3
Population: mITT Population. Only participants with data for primary successful electric cardioversion at the indicated timepoint were analyzed.
Measure: Number; unit: participants
Arm/Group | Fondaparinux | UFH/VKA
Number analyzed (Participants) | 151 | 148
participants | 137 | 133

8. Secondary Outcome: Number of Participants With a Thrombus in the Left Atrium (LA) or in the Left Atrial Appendage (LAA) at the Time of the Second TEE
Description: Atrial fibrillation (AF) causes stagnant blood in the LA or LAA and can lead to a thromboembolism. Stasis in the LAA represents the principal mechanism of thrombus formation in AF.
Time Frame: At second TEE (at Day 28+/-4)
Population: mITT Population. Only clot-positive participants at the time of the first TEE were analyzed.
Measure: Number; unit: participants
Arm/Group | Fondaparinux | UFH/VKA
Number analyzed (Participants) | 14 | 14
participants | 3 | 7

9. Secondary Outcome: Number of Thrombus-negative and Thrombus-positive Participants With Conversion to Sinus Rhythm
Description: Sinus rhythm is the normal beating of the heart, as measured by an ECG. Normal sinus rhythm not only indicates that the rhythm is normally generated by the sinus node and is traveling in a normal fashion in the heart, but it also indicates that the heart rate (the rate at which the sinus node is generating impulses) is within normal limits.
Time Frame: Baseline (Day 1) until Day 64 (4 days after the EOT [i.e., last administration of study drug]) for CP participants; Baseline until Day 36 (4 days after the EOT) for CN participants; and from Day 64 until the follow-up visit (FU) (Day 90+/-7)
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Fondaparinux | UFH/VKA
Number analyzed (Participants) | 174 | 170
participants
  Clot-negative par. until 4 days after EOT | 109 | 115
  Clot-positive par. until 4 days after EOT | 5 | 4
  Clot-negative participants until the FU | 105 | 106
  Clot-positive participants until the FU | 4 | 5

10. Secondary Outcome: Number of Participants Who Were Re-hospitalized
Description: Hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or out-patient setting. Re-hospitalization refers to an event of hospitalization after discharge for the initial hospitilization for the cardioversion.
Time Frame: as for outcome 2
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Fondaparinux | UFH/VKA
Number analyzed (Participants) | 174 | 170
participants
  until 4 days after EOT | 14 | 7
  until the FU | 18 | 11

ADVERSE EVENTS:
Time Frame: Participants were analyzed for the period from randomization up to the last administration of study treatment plus four days (up to Day 56+/-4 days).
Description: Serious adverse events (SAEs) and non-serious AEs were collected in members of the Safety Population, comprised of all participants included in the study, who had any post-baseline value, and who received at least one dose of study medication.
Arm/Group | Fondaparinux | UFH/VKA
Serious Adverse Events (participants affected / at risk) | 30/174 | 26/170
Other Adverse Events (participants affected / at risk) | 68/174 | 70/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux (N=174) | UFH/VKA (N=170)
Atrial fibrillation (Cardiac disorders) | 12 | 5
Cardiac failure (Cardiac disorders) | 4 | 3
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 2
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Ischemic cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Sinoatrial block (Cardiac disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Erosive esophagitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Death (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux (N=174) | UFH/VKA (N=170)
Atrial fibrillation (Cardiac disorders) | 13 | 11
Bradycardia (Cardiac disorders) | 2 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Intestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Edema (General disorders) | 4 | 3
Chest pain (General disorders) | 4 | 2
Edema peripheral (General disorders) | 1 | 3
Chest discomfort (General disorders) | 0 | 3
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Vessel puncture site hematoma (General disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 3
Hematoma (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 4 | 0
Hypertensive crisis (Vascular disorders) | 0 | 2
Phlebitis (Vascular disorders) | 2 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Sebaceous gland infection (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 2
Gout (Metabolism and nutrition disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 0
Dizziness (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 1 | 2
Disorientation (Psychiatric disorders) | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1
Transient psychosis (Psychiatric disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 5 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
International normalised ratio decreased (Investigations) | 0 | 1
International normalized ratio increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Skin operation (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.